CLINICAL TRIAL: NCT04752397
Title: The Influence of Extracorporeal Photopheresis on Skin Sclerosis - an Exploratory Clinical Study
Brief Title: The Influence of Extracorporeal Photopheresis on Skin Sclerosis
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Ulrike Blume-Peytavi, MD, Prof. Dr. Ulrike Blume-Peytavi, Charite University, Berlin, Germany
Other Study IDs: CRC-A-34
Record Dates: First submitted 2021-02-09; First posted 2021-02-12 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Scleroderma, Systemic; Graft Vs Host Disease; Eosinophilic Fasciitis; Morphea; Skin Sclerosis
Keywords: Extracorporeal photopheresis; Systemic Sclerosis; Morphea; Graft Vs Host Disease; Eosinophilic Fasciitis; Transepidermal water loss; Stratum corneum hydration; Skin firmness; High frequency ultrasonography; Skin surface sebum; Skin thickness; Biomarkers
MeSH Terms: conditions — Scleroderma, Systemic; Graft vs Host Disease; Eosinophilic Fasciitis; Scleroderma, Localized

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: None Retained — Blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Extracorporeal photopheresis (ECP), also known as extracorporeal photoimmunotherapy or photochemotherapy, is a leukapheresis-based therapy that has been in clinical use for over three decades after receiving FDA approval in 1988. Extracorporeal photopheresis was initially used for the treatment of T-cell lymphoma. Since its introduction, indications for initiating ECP were continuously extended to the treatment of Graft-versus-Host Disease (GvHD), systemic sclerosis, and in the field of solid organ transplantation. There is also evidence supporting the use of ECP in generalized morphea, a form of scleroderma limited to the skin, and in eosinophilic fasciitis, which is a rare, localized fibrosing disorder of the fascia.

Concluding the results of the published studies, there is evidence that ECP has a positive effect on fibrosing disorders of the skin. Furthermore, in clinical practice, it has been observed that patients with systemic sclerosis, who undergo ECP treatment, show improvement of the skin lesions or a deceleration in the formation progress of such lesions during the therapy. Same findings can be observed in patients with sclerotic skin lesions of the skin, for example in the context of a GvHD.

There are no clinical studies so far that describe these processes using objective measuring methods. Furthermore, the mechanism of action of ECP in systemic sclerosis and other fibrosing disorders with skin manifestations, has not yet been conclusively clarified. Serological markers for monitoring the progress of the therapy and determining the prognosis are also missing. Thus, a consensus regarding the frequency and duration of ECP for the therapy of systemic scleroderma or sclerotic diseases has not yet been reached.

This study aims at evaluating the influence of Extracorporeal Photopheresis on the quality and functionality of sclerotic skin lesions assessed by several objective methods. Furthermore, potential biomarkers, which are being investigated in current studies, are to be determined in order to evaluate the influence of ECP on those biomarkers and better understand the mechanism of action of ECP on systemic sclerosis and fibrosing disorders involving the skin.

DETAILED DESCRIPTION:
Background and Rationale:

Extracorporeal photopheresis:

In this immunomodulatory therapy, the apheresis leukocytes of the patients are irradiated with ultraviolet (UV) A in the presence of a photosensitizing agent, 8-methoxypsoralen prior to reinfusion to the patient. The mechanism of action of ECP has not yet been conclusively clarified. However, it has been shown that ECP modulates dendritic cells, modifies the cytokine profile and stimulates several T cell subpopulations, in particular regulatory T cells (Treg). The accumulated experience shows ECP to be well tolerated, with no clinically significant side effects and no long-term complications. Extracorporeal photopheresis is available as first-line as well as second-line therapy and can be combined with systemic drug therapies.

Scleroderma and ECP:

Scleroderma comprises a spectrum of autoimmune fibrosing disorders characterized by vascular alterations, fibrosis, and subsequent atrophy of the skin, subcutaneous tissue and muscles. Depending on the form of the disease, internal organs may also be affected in various degrees (e.g. alimentary tract, lungs, heart, kidney, central nervous system). It is usually classified into systemic sclerosis (generalized scleroderma) and morphea (localized scleroderma), distinguished by visceral involvement in the generalized form and disease limited to the skin and subcutaneous tissue in the localized form. Prognosis depends mainly on renal, cardiac and pulmonary manifestations.

The pathogenesis of scleroderma is not well understood. However, it is assumed that there is an initial damage to endothelial cells, a subsequent inflammatory reaction in which mainly T-lymphocytes, macrophages and mast cells are pathologically altered, and an activation of fibroblasts causing increased and disturbed collagen production, which finally leads to fibrosis. In addition, alterations in the innate and acquired immune response, a disturbed microcirculation and fibroblast dysfunction are also involved.

The therapy of patients with scleroderma is very limited. It is based on immunosuppression, which includes systemic steroids, azathioprine, cyclophosphamide, methotrexate, mycophenolate mofetil or interferons. Phototherapy is also a major component in the treatment of Scleroderma and ranges from narrowband to broadband UVB, UVA, UVA1, Psoralen-UVA (PUVA), and ECP. The key advantage of ECP for the treatment of scleroderma is the improvement of its skin manifestations. Nevertheless, there is also emerging evidence that suggests that ECP may play a role improving oral aperture size, joint mobility, skin ulcers and functional status. Furthermore, in contrast to the available immunosuppressive therapies, ECP has a low side effect profile. Τhe European Dermatology Forum recommends ECP as a second-line therapy or as part of adjuvant therapy in patients with scleroderma. There is currently no consensus on the duration and frequency of ECP for the treatment of scleroderma.

Graft-versus-Host Disease and ECP:

Graft-versus-host disease is a complex multiorgan disease, which can occur as a complication following allogeneic stem cell transplantation. Involvement of the skin represents the most common appearance of GvHD. According to the Consensus of National Institute of health further sub-classification can be done into acute and chronic GvHD.Corticosteroids are first-line therapy for both acute and chronic GvHD but due to its significant toxicity and an increasing number of patients developing steroid-refractory disease, many rescue therapies are currently available. ECP is a widely recommended treatment approach as a second-line treatment, especially in steroid refractory form of GvHD.

Eosinophilic fasciitis and ECP:

Eosinophilic fasciitis is a rare sclerodermiform syndrome of unknown etiology, characterized by the fibrosis of the muscular fascia and subcutaneous tissue accompanied with infiltration of eosinophils. There is little data regarding ECP in Eosinophilic fasciitis, however ECP may be beneficial.

Objectives:

The aim of this study is to investigate the influence of ECP on patients with autoimmune fibrosing disorders, including systemic sclerosis, morphea, sclerodermiform GvHD and eosinophilic fasciitis. More specifically, the following topics are going to be investigated:

1. Quality and functionality of skin lesions:

   1. Examination of lesional and clinically uninvolved skin during ECP treatment, using clinical evaluation and skin functional parameters. If possible, the examinations will take place before the initiation and during the ECP treatment. This depends on the stage of therapy of the participants, at the time they get included in the study.
   2. Evaluation of the influence of the frequency and the duration of ECP on the progress of the disease.
2. Alteration of biomarkers during the ECP treatment:

   1. Observation of specific potential biomarkers during the treatment in order to understand the mechanism of action of ECP as well as its influence in those biomarkers.
   2. Evaluation of biomarkers as possible prognostic markers.

Study design:

Prospective, monocentric, exploratory study with a single group of 10 subjects. Ten patients with sclerotic skin lesions due to systemic sclerosis, or morphea, or sclerodermiform GvHD or eosinophilic fasciitis will be enrolled in this clinical study. Subjects not having started first ECP treatment yet will be preferred for inclusion. The modified Rodnan skin score is widely accepted as a validated method to evaluate skin sclerosis, therefore its results will be considered as the primary outcome in this study. The study will include 8 visits for each included patient:

Screening visit, between week -2 and week 0

Baseline/inclusion visit, week 0

Intermediate visits, every 4 weeks ± 2

End of study visit, week 24± 2

Study setting:

The study will be conducted by the Clinical Research Center for Hair and Skin Science, Department of Dermatology and Allergy, Charité - Universitätsmedizin Berlin.

Patients with systemic sclerosis or sclerotic skin lesions who already receive or are planned to receive ECP treatment will be recruited in this study. In other words, they will receive the treatment regardless of their inclusion in the study. Normally, a 3-day inpatient stay in the clinic is required for a cycle of ECP treatment. The study visits will be carried out during this inpatient stay at the Department of Dermatology and Allergy, Charité - Universitätsmedizin Berlin. If necessary, additional appointments with the subjects will be made in the same setting.

Recruitment strategies:

Patients who receive ECP in the Department of Dermatology, Venerology and Allergology - Charité - Universitätsmedizin Berlin will be informed about the study by the study investigators.

Data collection methods:

1. Demographic data, medical history: An extended interview of the patient on his demographics, medical history, treatments and medications will be performed by an investigator during the inclusion visit.
2. Modified Rodnan skin score: The modified Rodnan skin score is a validated method to evaluate skin thickening in SSc worldwide.It will be performed by an investigator.
3. Skin physiological and functional parameters: Skin functional parameters will be determined at the uninvolved skin of the volar forearm or the gluteal area (control) and at one lesional skin area (target lesion), which may differ among the subjects but preferably would be in a contralateral area to the uninvolved skin area chosen. Before measurements are performed, subjects will rest for 30 minutes in a room with controlled environmental conditions (room temperature 22 °C± 2 °C; relative humidity 50% ± 10%) for acclimatization. The skin of the investigational sites must be open to air.

   Following parameters will be determined:

   Stratum corneum hydration (SCH): SCH will be measured using the Corneometer CM 825 (Courage + Khazaka, Colonge, Germany), which measures the hydration level of the stratum corneum as electrical capacitance. The measurement is based on the differences of the dielectric constant of water and other substances. The arbitrary units range from 0 to 120, higher readings indicate higher stratum corneum hydration.

   Transepidermal water loss (TEWL): TEWL will be measured using the Tewameter TM 300 (Courage + Khazaka, Colonge, Germany). The probe of the instrument measures the density gradient of the water evaporation from the skin indirectly by the two pairs of sensors (temperature and relative humidity) inside the hollow cylinder. Water evaporation is captured in gram per hour per m². Higher values indicate a higher transepidermal water loss.

   Skin firmness: A Cutometer Dual MPA 580 (Courage + Khazaka, Colonge, Germany) will be used. The instrument measures skin deformation after repeated cycles of suction and release. The resistance of the skin to the negative pressure and its ability to return into its original position are displayed as curves (penetration depth in mm/time) in real time during the measurement.

   Skin surface sebum level: A Sebumeter SM 815 (Courage + Khazaka, Colonge, Germany) will be used. The measurement is based on grease spot photometry. The measurement cassette contains a special tape that becomes transparent when it comes into contact with sebum on the surface of the skin. In order to make a measurement the cassette is inserted into an aperture on the device where the transparency of the tape is measured. The transparency is measured by sending light through the tape, using a light source in the aperture. The light is reflected by a mirror behind the tape and a photocell measures the transparency. The change in the amount of light transmission represents the sebum content of the tape, which is displayed in units from 0-350. Higher values indicate a higher lipid level.

   Skin thickness: A Dermascan C ultrasound scanner (Cortex Technology, Denmark) with a 20MHz probe will be used.
4. Biomarkers: Biomarkers will be determined via blood sampling. Two CPDa tubes and two serum tubes will be used at each blood collection. Blood samples will be collected at three time-points during an inpatient stay; immediately before the start of ECP on day one, immediately after the ECP treatment on day one and at the patient's discharge on day three. Serum levels of specific cytokines and chemokines will be determined using ELISA. Percentage counts of specific T-cell subpopulations will be obtained by fluorescence-activated cell sorting analysis (FACS), using the following surface markers: CD3, CD4, CD45RA, CD127, CD25, CXCR3, CXCR5 and CCR6.

Data management:

A paper source data will be created for this study. Data including demographics, medical history, measurement results and clinical score results will be completed during the study visits in written form. Data from the source data will be extracted and entered into a data file by the data manager using the software IBM SPSS Statistics 26. The database will be stored on a secured digital server of the Charité - Universitätsmedizin Berlin.

Statistical methods:

Descriptive comparative statistical analysis will be conducted. All parameters will be described using measures of central tendency and measures of variability or dispersion. This is an exploratory study therefore a formal sample size calculation is not planned.

Monitoring:

Data Monitoring: Planned.

Harms: The participants will not be monitored for adverse events because the study is considered as non-interventional. All subjects will receive ECP treatment regardless of their inclusion in this study. Furthermore, all non-invasive measurements as well as the blood sampling will be conducted during the subjects' planned hospitalization.

Auditing: Not planned.

ELIGIBILITY:
Inclusion Criteria:

1. Systemic sclerosis, morphea, sclerodermiform GvHD or eosinophilic fasciitis, with duration less than 5 years.
2. Ability and willingness to both understand and carry out the study requirements

Exclusion Criteria:

1. Participation in another study, currently or in the previous four weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who receive ECP in the Clinic of Dermatology, Venerology and Allergology - Charité - Universitätsmedizin Berlin.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2021-02-12 (Actual); Primary Completion 2021-08-17 (Actual); Study Completion 2021-09-06 (Actual)

PRIMARY OUTCOMES:
Modified Rodnan Skin score | Week 4 ± 2
  The skin thickening is being assessed by palpation of the skin in 17 areas of the body using a 0-3 scale, where 0 = normal, 1 = mild thickness, 2 = moderate thickness and 3 = severe thickness (total score=51).
Modified Rodnan Skin score | Week 8 ± 2
  The skin thickening is being assessed by palpation of the skin in 17 areas of the body using a 0-3 scale, where 0 = normal, 1 = mild thickness, 2 = moderate thickness and 3 = severe thickness (total score=51).
Modified Rodnan Skin score | Week 12 ± 2
  The skin thickening is being assessed by palpation of the skin in 17 areas of the body using a 0-3 scale, where 0 = normal, 1 = mild thickness, 2 = moderate thickness and 3 = severe thickness (total score=51).
Modified Rodnan Skin score | Week 16 ± 2
  The skin thickening is being assessed by palpation of the skin in 17 areas of the body using a 0-3 scale, where 0 = normal, 1 = mild thickness, 2 = moderate thickness and 3 = severe thickness (total score=51),
Modified Rodnan Skin score | Week 20 ± 2
  The skin thickening is being assessed by palpation of the skin in 17 areas of the body using a 0-3 scale, where 0 = normal, 1 = mild thickness, 2 = moderate thickness and 3 = severe thickness (total score=51).
Modified Rodnan Skin score | Week 24 ± 2
  The skin thickening is being assessed by palpation of the skin in 17 areas of the body using a 0-3 scale, where 0 = normal, 1 = mild thickness, 2 = moderate thickness and 3 = severe thickness (total score=51).

SECONDARY OUTCOMES:
Skin thickness at control skin area | Week 12 ± 2
  Means of triplicate measurements in millimetres (mm).
Skin thickness at lesional skin area | Week 12 ± 2
  Means of triplicate measurements in mm.
Skin thickness at control skin area | Week 24 ± 2
  Means of triplicate measurements in mm.
Skin thickness at lesional skin area | Week 24 ± 2
  Means of triplicate measurements in mm.
Transepidermal water loss (TEWL) at control skin area | Week 12 ± 2
  Means of triplicate measurements in g/m²/h.
TEWL at lesional skin area | Week 12 ± 2
  Means of triplicate measurements in g/m²/h.
TEWL at control skin area | Week 24 ± 2
  Means of triplicate measurements in g/m²/h.
TEWL at lesional skin area | Week 24 ± 2
  Means of triplicate measurements in g/m²/h.
Stratum corneum hydration (SCH) at control skin area | Week 12 ± 2
  Means of triplicate measurements in arbitrary units (0-120).
SCH at lesional skin area | Week 12 ± 2
  Means of triplicate measurements in arbitrary units (0-120).
SCH at control skin area | Week 24 ± 2
  Means of triplicate measurements in arbitrary units (0-120).
SCH at lesional skin area | Week 24 ± 2
  Means of triplicate measurements in arbitrary units (0-120).
Skin firmness at control skin area | Week 12 ± 2
  The final deformation (Uf) will be determined. Means of triplicate measurements in mm.
Skin firmness at lesional skin area | Week 12 ± 2
  The final deformation (Uf) will be determined. Means of triplicate measurements in mm.
Skin firmness at control skin area | Week 24 ± 2
  The final deformation (Uf) will be determined. Means of triplicate measurements in mm.
Skin firmness at lesional skin area | Week 24 ± 2
  The final deformation (Uf) will be determined. Means of triplicate measurements in mm.
Skin surface sebum level at control skin area | Week 12 ± 2
  Means of triplicate measurements in arbitrary units (0-350).
Skin surface sebum level at lesional skin area | Week 12 ± 2
  Means of triplicate measurements in arbitrary units (0-350).
Skin surface sebum level at control skin area | Week 24 ± 2
  Means of triplicate measurements in arbitrary units (0-350).
Skin surface sebum level at lesional skin area | Week 24 ± 2
  Means of triplicate measurements in arbitrary units (0-350).
Serum levels of proinflammatory factors Interleukin 4 (IL-4), Interleukin 9 (IL-9), Interleukin 33 (IL-33) and Transforming growth factor beta (TGF-beta). | Week 8 ± 2
  pg/ml at time point 3 (after completion of the cycle).
Serum levels of Platelet factor 4 (CXCL4). | Week 8 ± 2
  pg/ml at time point 3.
Acute change in serum levels of proinflammatory factors IL-4, IL-9, IL-33 and TGF-beta. | Week 8 ± 2
  pg/ml. Change in serum levels between time point 1(before the start of the ECP treatment on day one) and time point 2 (immediately after the ECP treatment on day one).
Acute change in serum levels of Platelet factor 4 (CXCL4). | Week 8 ± 2
  pg/ml. Change in serum levels between time point 1 and time point 2.
Change in serum levels of proinflammatory factors IL-4, IL-9, IL-33 and TGF-beta after ECP cycle. | Week 8 ± 2
  pg/ml. Change in serum levels between time point 1 and time point 3.
Change in serum levels of CXCL4 after ECP cycle. | Week 8 ± 2
  pg/ml. Change in serum levels between time point 1 and time point 3.
Serum levels of proinflammatory factors IL-4, IL-9, IL-33 and TGF-beta. | Week 16 ± 2
  pg/ml at time point 3.
Serum levels of CXCL4. | Week 16 ± 2
  pg/ml at time point 3.
Acute change in serum levels of proinflammatory factors IL-4, IL-9, IL-33 and TGF-beta. | Week 16 ± 2
  pg/ml. Change in serum levels between time point 1 and time point 2.
Acute change in serum levels of CXCL4. | Week 16 ± 2
  pg/ml. Change in serum levels between time point 1 and time point 2.
Change in serum levels of proinflammatory factors IL-4, IL-9, IL-33 and TGF-beta after ECP cycle | Week 16 ± 2
  pg/ml. Change in serum levels between time point 1 and time point 3.
Change in serum levels of CXCL4 after ECP cycle. | Week 16 ± 2
  pg/ml. Change in serum levels between time point 1 and time point 3.
Serum levels of proinflammatory factors IL-4, IL-9, IL-33 and TGF-beta. | Week 24 ± 2
  pg/ml at time point 3.
Serum levels of CXCL4. | Week 24 ± 2
  pg/ml at time point 3.
Acute change in serum levels of proinflammatory factors IL-4, IL-9, IL-33 and TGF-beta. | Week 24 ± 2
  pg/ml. Change in serum levels between time point 1 and time point 2.
Acute change in serum levels of CXCL4. | Week 24 ± 2
  pg/ml. Change in serum levels between time point 1 and time point 2.
Change in serum levels of proinflammatory factors IL-4, IL-9, IL-33 and TGF-beta after ECP cycle. | Week 24 ± 2
  pg/ml. Change in serum levels between time point 1 and time point 3.
Change in serum levels of CXCL after ECP cycle. | Week 24 ± 2
  pg/ml. Change in serum levels between time point 1 and time point 3.
Percentage counts of T helper type 1 (Th1), T helper type 2 (Th2), T helper type 17 (Th17) and Treg cells. | Week 8 ± 2
  Percentage (%) at time point 3.
Acute change in percentage counts of Th1, Th2, Th17 and Treg cells | Week 8 ± 2
  Percentage (%). Change between time point 1 and time point 2.
Change in percentage counts of Th1, Th2, Th17 and Treg cells after ECP cycle. | Week 8 ± 2
  Percentage (%). Change between time point 1 and time point 3.
Percentage counts of Th1, Th2, Th17 and Treg cells. | Week 16 ± 2
  Percentage (%) at time point 3.
Acute change in percentage counts of Th1, Th2, Th17 and Treg cells. | Week 16 ± 2
  Percentage (%). Change between time point 1 and time point 2.
Change in percentage counts of Th1, Th2, Th17 and Treg cells after ECP cycle. | Week 16 ± 2
  Percentage (%). Change between time point 1 and time point 3.
Percentage counts of Th1, Th2, Th17 and Treg cells. | Week 24 ± 2
  Percentage (%) at time point 3.
Acute change in percentage counts of Th1, Th2, Th17 and Treg cells. | Week 24 ± 2
  Percentage (%). Change between time point 1 and time point 2.
Change in percentage counts of Th1, Th2, Th17 and Treg cells after ECP cycle. | Week 24 ± 2
  Percentage (%). Change between time point 1 and time point 3.

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Blume-Peytavi, Prof. MD, Principal Investigator — ulrike.blume-peytavi@charite.de
Locations (1):
- Charité-Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cho A, Jantschitsch C, Knobler R. Extracorporeal Photopheresis-An Overview. Front Med (Lausanne). 2018 Aug 27;5:236. doi: 10.3389/fmed.2018.00236. eCollection 2018. PMID 30211164
- [Background] Zhou XA, Choi J. Photopheresis: Advances and Use in Systemic Sclerosis. Curr Rheumatol Rep. 2017 Jun;19(6):31. doi: 10.1007/s11926-017-0662-8. PMID 28466383
- [Background] Knobler R, Berlin G, Calzavara-Pinton P, Greinix H, Jaksch P, Laroche L, Ludvigsson J, Quaglino P, Reinisch W, Scarisbrick J, Schwarz T, Wolf P, Arenberger P, Assaf C, Bagot M, Barr M, Bohbot A, Bruckner-Tuderman L, Dreno B, Enk A, French L, Gniadecki R, Gollnick H, Hertl M, Jantschitsch C, Jung A, Just U, Klemke CD, Lippert U, Luger T, Papadavid E, Pehamberger H, Ranki A, Stadler R, Sterry W, Wolf IH, Worm M, Zic J, Zouboulis CC, Hillen U. Guidelines on the use of extracorporeal photopheresis. J Eur Acad Dermatol Venereol. 2014 Jan;28 Suppl 1(Suppl 1):1-37. doi: 10.1111/jdv.12311. PMID 24354653
- [Background] Hassani J, Feldman SR. Phototherapy in Scleroderma. Dermatol Ther (Heidelb). 2016 Dec;6(4):519-553. doi: 10.1007/s13555-016-0136-3. Epub 2016 Aug 12. PMID 27519050
- [Background] Gabrielli A, Avvedimento EV, Krieg T. Scleroderma. N Engl J Med. 2009 May 7;360(19):1989-2003. doi: 10.1056/NEJMra0806188. No abstract available. PMID 19420368
- [Background] Guggino G, Lo Pizzo M, Di Liberto D, Rizzo A, Cipriani P, Ruscitti P, Candore G, Gambino CM, Sireci G, Dieli F, Giacomelli R, Triolo G, Ciccia F. Interleukin-9 over-expression and T helper 9 polarization in systemic sclerosis patients. Clin Exp Immunol. 2017 Nov;190(2):208-216. doi: 10.1111/cei.13009. Epub 2017 Aug 23. PMID 28681919
- [Background] Li L, Zhu H, Zuo X. Interleukin-33 in Systemic Sclerosis: Expression and Pathogenesis. Front Immunol. 2018 Nov 15;9:2663. doi: 10.3389/fimmu.2018.02663. eCollection 2018. PMID 30498500
- [Background] Sacchetti C, Bai Y, Stanford SM, Di Benedetto P, Cipriani P, Santelli E, Piera-Velazquez S, Chernitskiy V, Kiosses WB, Ceponis A, Kaestner KH, Boin F, Jimenez SA, Giacomelli R, Zhang ZY, Bottini N. PTP4A1 promotes TGFbeta signaling and fibrosis in systemic sclerosis. Nat Commun. 2017 Oct 20;8(1):1060. doi: 10.1038/s41467-017-01168-1. PMID 29057934
- [Background] Matsushita T, Takehara K. An update on biomarker discovery and use in systemic sclerosis. Expert Rev Mol Diagn. 2017 Sep;17(9):823-833. doi: 10.1080/14737159.2017.1356722. Epub 2017 Jul 25. PMID 28730919
- [Background] Romano C, Rubegni P, De Aloe G, Stanghellini E, D'Ascenzo G, Andreassi L, Fimiani M. Extracorporeal photochemotherapy in the treatment of eosinophilic fasciitis. J Eur Acad Dermatol Venereol. 2003 Jan;17(1):10-3. doi: 10.1046/j.1468-3083.2003.00587.x. PMID 12602960
- [Background] Abraham DJ, Krieg T, Distler J, Distler O. Overview of pathogenesis of systemic sclerosis. Rheumatology (Oxford). 2009 Jun;48 Suppl 3:iii3-7. doi: 10.1093/rheumatology/ken481. PMID 19487220